CLINICAL TRIAL: NCT04367194
Title: Objective Examination and Rehabilitation Treatment of Patients With BPPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somogy Megyei Kaposi Mór Teaching Hospital (Other)
Responsible Party: Principal Investigator, Tollár József, Principal Investigator, Somogy Megyei Kaposi Mór Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IKEB2019/15
Record Dates: First submitted 2020-04-23; First posted 2020-04-29 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Postural Vertigo; Vertigo, Paroxysmal; Vertigo, Positional; Coordination Disorder, Developmental; Coordination and Balance Disturbances
Keywords: vertigo; balance; instability; rehabilitation
MeSH Terms: conditions — Vertigo; Motor Skills Disorders | interventions — Neurological Rehabilitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BPPV intervention (Experimental): After examination of the patients, the patients undergo neurorehabilitation. We use virtual reality therapy. Patients perform a submaximal load that is monitored by a polar clock. We develop endurance, coordination, sensory integration, visual and acoustic input, vestibular training, proprioception training.
  Interventions: Behavioral: Neurorehabilitation
- BPPV Epley (Experimental): Only Epley training.
  Interventions: Behavioral: Neurorehabilitation
- BPPV Optocinetic (Experimental): Only Optocinetic training.
  Interventions: Behavioral: Neurorehabilitation

INTERVENTIONS:
Behavioral: Neurorehabilitation — After examination of the patients, the patients undergo neurorehabilitation. We use virtual reality therapy. Patients perform a submaximal load that is monitored by a polar clock. We develop endurance, coordination, sensory integration, visual and acoustic input, vestibular training, proprioception training.
  Other Names: BPPV group

SUMMARY:
Dizziness (BPPV) causes severe deterioration in quality of life, incoordination, and instability.

In the study, we selected a minimum of 100 patients with BPPV who were examined after specialist care. After the acute phase, a physical survey is performed where movement and coordination are examined.

After the results, the patients undergo a rehabilitation training. The workout is submaximal and high intensity that is done for 3 weeks.

Hypothesis: As a result of training, it is possible that the remaining feeling of dizziness and insecurity, impaired coordination will decrease or disappear.

ELIGIBILITY:
Inclusion Criteria:

* For a patient with BPPV
* With a lack of coordination
* Dizziness
* Ear nose laryngeal examination
* Neurological examination

Exclusion Criteria:

* other neurological diseases
* cardiological diseases
* underwent surgery
* severe joint pain
* alcoholism
* dementia
* drug

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
EQ5D-5L | 5 weeks
  Quality of life testing is taken with a test. The therapist scores the answers to the questions asked on a scale. The end result determines the quality of life.
Beam Walking test | 5 weeks
  The patient walks on slats of varying width. During the examination, the therapist says the tasks (Eg: counting backwards). The study detects the determination of dynamic equilibrium.
Posturography | 5 weeks
  Noninvasive intervention where static equilibrium is examined. The program determines the quality and frequency of the displacements.

CONTACTS AND LOCATIONS:
Locations (1):
- Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár, Somogy County, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BPPV rehabilitation — https://www.ncbi.nlm.nih.gov/pubmed/?term=BPPV+rehabilitation